| Ir | <b>rvesti</b> | gation of | the Effective | veness of <b>V</b> | Visual Feedb | oack |
|---|---|---|---|---|---|---|
| Trai | ning | on Uppei | Extremity | Functions | s in Cerebra | l Palsy |

Study Protocol with Statistical Analysis Plan (SAP) and Informed Consent Form (ICF)

# Investigation of the Effectiveness of Visual Feedback Training on Upper Extremity Functions in Cerebral Palsy

**Study Protocol** 

(Pages 2-6)

#### **Study Protocol**

Study titled 'Investigation of the Effectiveness of Visual Feedback Training on Upper Extremity Functions in Cerebral Palsy was approved by Marmara University Faculty of Medicine Clinical Researches Ethics Committee meeting on 05.01.2018 with approval number: 09.2018.007 (Annex-1).

The legal representatives of the children who participated in the study were informed about the aim, duration and the programs to be applied throughout the study. Volunteer Information Form has been signed and approved in accordance with the standards deemed appropriate by the Clinical Researches Ethics Committee of Marmara University Faculty of Medicine (This form can be seen on Informed Consent Form (ICF) section). The study was conducted in accordance with the Declaration of Helsinki.

### **Hypothesis of the Study**

H0: Addition of the exercises performed with Cogniboard® Light Trainer device to the neurodevelopmental (NDT) based rehabilitation program in patients with cerebral palsy does not contribute positively in improving the efficiency of upper extremity functions.

H1: Addition of the exercises performed with Cogniboard® Light Trainer device to the neurodevelopmental (NDT) based rehabilitation program in patients with cerebral palsy contributes positively to improve the efficiency of upper extremity functions.

### Randomization of the Study Groups

Children with Cerebral Palsy who applied to the Dilbade Education and Rehabilitation Center for rehabilitation were invited to participate to the study. Children who volunteered to participate and whom met the criteria for participation were randomized with simple random sampling method and divided into two groups. Individual Neurodevelopmental (NDT) based rehabilitation programs were applied to the participants in both groups. The Cogniboard® Light Trainer education system was added to the rehabilitation program of the Group II (the study group).

#### **Inclusion Criteria**

- Volunteered to participte,
- The child and the family have agreed to participate in the study,
- Having a diagnosis of Cerebral Palsy,
- Children aged between 4 18 years,
- Having upper extremity spasticity (0), (1), (1+) according to the modified Ashworth Scale (MAS)
- To be able to cooperate to the exercises

#### **Exclusion Criteria**

- Botulinum Toxin (BOTOX) injection applied to the upper extremity within the last 6 months,
- Congenital deformity in upper extremity
- Epileptic attack history,
- Any cardiac or orthopedic problem,
- Visual or hearing impairement

### **Applied Evaluations**

Evaluations are applied twice: before and after the study. All evaluation data are noted to 'Participants Tracking Form' (Annex-2). Spasticity was defined with 'Modified Ashworth Scale'; upper extremity joint range of motion (ROM) with 'goniometer'; grip and pinch strength with 'dynamometer'; hand skills with 'Minnesota Hand Skill Test'; functional abilities with 'Childhood Health Assessment Questionnaire (CHAQ) and functional level with 'Gross Motor Function Classification System (GMFCS)'

### **Treatment Program**

The participants in our study were all rehabilitated in Dilbade Education and Rehabilitation Center twice a week for 8 weeks, a total of 16 sessions (Duration of one session is 45 minutes).

Group I (Control Group) received individual Neurodevelopmental (NDT) based rehabilitation program.

Group II (Study Group) received individual NDT based rehabilitation program (35 minutes) + Cogniboard® Light Trainer education (10 minutes).

### Cogniboard® Light Trainer Education Protocol

Upper limb exercises were applied to the study group with the device which is a training program with visual feedback for 10 minutes in addition to individual 35 minutes neurodevelopmental treatment program. Devices were placed in the mirror so that the participants could see their own reflection. The distances of the participants to the mirror were proportional to their height. For children between 100-149 cm, the distance of the child with the mirror was set as 40 cm and for the children between 149-175 cm, 50 cm. Eight devices were placed in the mirror within the reach of the participant. While the shoulder and wrist were flexed, the shoulder was placed in the lateral distances that the shoulder could reach while the shoulder was in 90°, while the shoulder was in extension and the other devices were placed between these points (Picture 1).



(Picture 1. Application of Cogniboard® Light Trainer Education Device)

### Neurodevelopmental Therapy (NDT) Based Upper Extremity Rehabilitation

In accordance with the needs of the patients for their gross motor functions, the children in both groups were included in the NDT program, which was determined according to the age, sex, mental status and preferences of the individual. NDT program included; rehabilitation of muscle tonus disorders, sensory-perception-motor integrity enhancement, exercises to increase upper extremity functions, stretching and strengthening exercises due to muscular shortness and weakness, exercises to accommodate movements in daily life, and training of activities such as standing up, eating, walking, body care.

# Investigation of the Effectiveness of Visual Feedback Training on Upper Extremity Functions in Cerebral Palsy

**Statistical Analysis Plan (SAP)** 

(Pages 7-8)

### **Statistical Analysis Plan (SAP)**

The statistical program Statistical Package for Social Sciences (SPSS) Version 11.5 (SPSS Inc., Chicago, IL, USA) was used in the data analysis of the study. The p value of p<0.05 was considered to be statistically significant in the data analysis. Shaphiro-Wilks test was used to investigate the appropriateness of the variables to normal distribution.

In the comparison of the nominal characteristics of the participants in both groups, such as gender, CP type, GMFCS and dominant side, Fisher Precise Chi-Square Test was used.

The initial demographic characteristics such as age, height, weight, body mass index (BMI) of the participants in both groups and the changes before and after the treatment were compared with Independent Samples t-Test and Paired Samples t-Test.

# Investigation of the Effectiveness of Visual Feedback Training on Upper Extremity Functions in Cerebral Palsy

**Informed Consent Form (ICF)** 

(Pages 9 - 13)

### **Informed Consent Form (ICF)**

### **Description of the Physiotherapist**

This study, if you accept your child to be participated, is a scientific research and it is titled as 'Investigation of the Effectiveness of Visual Feedback Training on Upper Extremity Functions in Cerebral Palsy'. In this study, individuals with Cerabral Palsy will be evaluated in terms of upper extremity (arm) functions, upper extremities' joint range of motion with universal goniometer, gripping force with dynamometer, pinching force with pinchmeter, spasticity will be defined with Modified Ashworth Scale (MAS), hand skills with 'Minnesota Hand Skill Test'; functional abilities with 'Childhood Health Assessment Questionnaire (CHAQ) and functional level with 'Gross Motor Function Classification System (GMFCS)'. The study, which is planned to last in 8 weeks, requires participants to attend the study regularly for 2 days a week and each day for one session which is 45 minutes. There will be no disruption of the body during the process.

This research will be carried out by Physiotherapist Dilara Merve SARI (Tel: 0533 344 46 01) and will be under the supervision of Assoc. Prof. Dr. Tuğba KURU ÇOLAK at Marmara University, Institute of Health Sciences, Department of Physiotherapy and Rehabilitation.

Your child is being invited to a research project. It is very important you to understand why and how this research will be done before making a decision. Please take some time and read the following informations carefully, discuss it with others if you wish. If you have an unclear section or need more detailed information, you can get information from us. You are invited to our research because we think your child matches the criterias to be included. We would like to note that participation is voluntary and that refusal to participate does not lead to any penalty or loss of any benefit. In the same way, you can withdraw from the research at any time.

After getting the demographic information of the participants, the upper extremity functions will be measured by the above physiotherapist and with the mentioned tests. The evaluation tests will be repeated 2 times throughout the treatment. The data obtained from the assessments will be recorded in the computer and the changes during pre- and post-treatment will be analyzed.

The assessments applied to the participants in our research do not have any known harm. In the event of any unexpected damage in the evaluation process or during the rehabilitation process, the information will be given immediately to you. In case of any damage to the participants, the necessary applications shall be covered by the researchers without any recourse. For this, you will not be charged any fees, neither you nor your social security insurance.

While participation in the research does not help you immediately, it is hoped that our research results will have benefits for the organization, society or science in the future. You will not be charged any fees for the purposes of the research or for the social security institution to which you are affiliated.

### **Consent of the Participant**

I have read the entire information form clearly and understood or because I do not know how to read/not able to or do not understand the language it was read or translated to me. I was given the opportunity to ask, evaluate and decide on my health status both during and after my application and when filling this form in. All kinds of treatment and diagnostic alternatives, including the possibility of not getting the treatment, their risks and dangers are explained.

Name and the Surname of the Participant and Legal Representative:

Date: Signature:

Name and Surname of the Withness:

Date: Signature:

### **Declaration of the Physiotherapist**

I gave the patient the necessary information about the study and the procedures to be performed. I believe that the patient understood this information, asked me the questions that she/he wanted to ask, and accepted the process with her/his free will.

Researcher: Physiotherapist Dilara Merve Sarı

Address: Dilbade Education and Rehabilitation Center – Silahtaraga, 129 34050 Eyup /

Istanbul / Turkey

Mobile Phone: +90 533 344 46 01 E-mail: dilaramervesari@gmail.com

Date: Signature:

### **Declaration of the Participant / Legal Representative**

Ms. Dilara Merve SARI stated that a medical research will be carried out and the above information about this research was explained to me. I know my child is invited to this research as a participant. If I participate in this research, I believe that the confidentiality of the information of my child during research will be treated with great care and respect. I was given enough information that my child's personal information would be protected with care during the use of the research and the results will only used for educational and scientific purposes. During the research I can withdraw my child from the study at any time without any cause (But in that case I am aware of the difficult situation it would cause to the reaseachers if I do not give any notice). I don't take any financial responsibility for the research expenses. There will be no payment for me. Whether directly, indirectly arised any health problem that may occur during the research, I will not undergo any monetary burden. When we encounter any health problem during the research; at any hour, I know I can call physiotherapist Dilara Merve SARI from +90 533 344 46 01 (mobile).

My child does not have to be participated in this research or may not participate. We have not experienced any compelling behavior to participate in the research. If we refuse to participate, I know that this will not bring any harm to our medical care and our relationship with my physiotherapist.

I have understood all the explanations made to me in detail. At the end of a certain period of thinking on my own, I decided that my child could take part in this research project as a participant. On behalf of my child, I accept this invitation voluntarily.

### **Voluntary Approval Form**

**Mobile Phone:** +90 533 344 46 01

Date:

I have read the text above which shows the information that should be given to the volunteer before investigating. These were written and was explained verbally. With these conditions, I agree to participate in this research without any pressure or compulsion on me and my child. A signed 2 copies of this form, which consists of 4 pages, a copy of the documents will be given to me.

| Name and the | Surname of the | Participant and | Legal Re | presentative: |
|---|---|---|---|---|
|---|---|---|---|---|

| Date: | Signature: |
|---|---|
| Name and Surname of the Withness (who have witnesse end): | ed the process of receipt until the |
| Date: | Signature: |
| The researcher who made the explanations, | |
| Researcher: Physiotherapist Dilara Merve Sarı | |
| Address: Dilbade Education and Rehabilitation Center – S | Silahtaraga, 129 34050 Eyup / |
| Istanbul / Turkey | |

**E-mail:** dilaramervesari@gmail.com

**Signature:** 

**Annex 1.** Marmara University Faculty of Medicine Clinical Researches Ethics Committee Approval (Approval made at the meeting on 05.01.2018 with number: 09.2018.007)



### Marmara Üniversitesi Tıp Fakültesi Klinik Araştırmalar Etik Kurulu

| | PROTOKOL KODU | 09.2018.007 |
|---|---|---|
| BAŞVURU<br>BİLGİLERİ | PROJE ADI | Serebral Palsili Olgularda Görsel Geri Bildirimli Eğitimin<br>Üst Ekstremite Fonksiyonlarına Etkinliğinin Araştırılması |
| BILGILERI | SORUMLU ARAŞTIRICI ÜNVANI/ADI | Doç. Dr. Tuğba KURU ÇOLAK |

| | Farih 05.01.2018<br>Yukarıda başvuru bilgileri veri | ilen araştırma başvuru dosyası ve | ilgili belgeler araştırı | manın gerekçe, amaç | , yaklaşım ve yöntemleri dikk |
|---|---|---|---|---|---|
| | ılınarak incelenmiş ve gerçekl<br>sonrasında yapılacak her türlü<br>onayının yenilenmesi gerekmek | eştirilmesinde sakınca bulunmadı<br>i proje değişiklikleri (katılımcılar<br>tedir. | gi için Kurulumuzca<br>, başlık vb.) veya pro | onaylanmasına oy bi<br>otokol değişikliklerini | n Etik Kurula bildirilerek p |
| YELER | | | | | |
| Unvani / Adı / Soyadı | Uzmanlık Dalı | Kurumu / EK Üyeliği | Onaylanan Proje<br>ile İlişkisi | Toplantiya<br>katılım | İmza |
| Prof.Dr. Haner DİRESKENEL | Romatoloji | M.Ü Tıp Fakültesi/ Başkan | Var Yok | Evet Hayır | of he |
| Prof.Dr. Tülin ERGUN | Dermatoloji | M.Ü Tıp Fakültesi/Başkan<br>Yrd. | <br>Var Yok | Evet Hayır | 1 |
| Prof. Dr. Şefik GÖRKEY | Tıp Tarihi ve Etik | M.Ü Tıp Fakültesi/Üye | <br>Var Yok | Evet Hayır | 1 Galey |
| Prof.Dr. Handan KAYA | Patoloji | M.Ü Tıp Fakültesi/Üye | <br>Var Yok | Evet Hayır | 3/ |
| Prof.Dr. M.Bahadır GÜLLÜÖÖ | GLU Genel Cerrahi | M.Ü Tıp Fakültesi/Üye | Var Yok | Evet Hayır | Juful- |
| Prof.Dr. Atila KARAALP | Farmakoloji | M.Ü Tıp Fakültesi/Üye | <br>Var Yok | EVET HAYIR | 1 MIN |
| Prof.Dr. Semra SARDAŞ | Eczacı | M.Ü Eczacılık Fak./Üye | <br>Var Yok | Evet Hayır | Tour |
| Prof.Dr. Başak DOĞAN | Diş Hekimi | M.Ü Diş Hekimliği Fak./Üye | <br>Var Yok | Evet Hayır | 1 |
| Prof. Dr. Beste Melek ATASOY | Radyasyon<br>Onkolojisi | M.Ü Tıp Fakültesi/Üye | Var Yok | Evet Hayır | |
| Doç. Dr. Elif KARAKOÇ AYDI | NER Çocuk Sağlığı ve<br>Hastalıkları | M.Ü Tıp Fakültesi/Üye | Var Yok | Evet Hayır | A. M. |
| Doç.Dr. Meltem KORAY | Diş Hekimi | İstanbul Üniv. Diş Hekimliği<br>Fak./Üye | Var Yok | Evet Hayır | M |
| Doç. Dr. Gürkan SERT | Hukukçu | M.Ü Tıp Fakültesi/Üye | Var Yok | Evet Hayır | 3 |
| Doç.Dr: Figen DEMİR | Halk Sağlığı | Acıbadem Üniv. Tıp Fak. | Var Yok | Evet Hayır | |
| Doç.Dr. Pınar Mega TİBER | Biyofizik | M.Ü Tıp Fakültesi/Üye | Var Yok | Evet Hayır | |
| Gözde Aynur MİRZA | Sağlık Mensubu<br>olmayan kişi | Serbest | Var Yok | Evet Hayır | qui |

## Annex 2. Participants Tracking Form

| Participant's Name - Surnam | ie: | | | |
|---|---|---|---|---|
| Legal Representative Name - | Surname: | | | |
| Phone number: | | | | |
| Age / Gender: | Height | : | Weig | ht: |
| Date of birth: | | | | |
| Type of Cerebral Palsy (CP) | (Mark X): | Spastic | Diskinetic | Ataxic |
| Which side of the arm is effec | cted mostly? | | | |
| Which side is your dominant | side? | | | |
| How did the problem occur? | (Preterm bi | rth, after bi | rth etc. Please o | explain.) |
| How many years have you be | en going to s | a rehahilitat | ion center? | |
| now many years have you be | on going to t | . i chabilitat | ion center. | |
| Did you have any operations? | ? Please writ | e if you did: | | |
| Are you using any device? If | so what aro | thoyt? | | |
| Are you using any device: It | so, what are | meyt. | | |
| Evaluations: | | | | |
| Muscle Tone: (According to t | he Modified | Ashworth S | Scale 0/1/1+/2/3 | 3/4) |
| | Right | or Left Arm | (Please mark) | |
| Hand Wrist Function: | | | | |
| Elbow Flexion: | | | | |
| Supination: | | | | |
| Do you have any additional m | nedical prob | lems? | | |
| Yes / What is it?: | _ | | | |
| No: | | | | |

| Range of Motion: | | Before Treatment | After Treatment |
|------------------|------------|------------------|-----------------|
| Chauldan | Flexion | | |
| Shoulder | Abduction | | |
| Elbow | Flexion | | |
| | Extension | | |
| Front Arm | Supination | | |
| | Pronation | | |
| Hand Wrist | Flexion | | |
| manu wrist | Extension | | |

| Muscle Strength | Before Treatment | After Treatment |
|-----------------|------------------|-----------------|
| Grasping | | |
| Tip Pinch | | |
| Lateral Pinch | | |
| Triple Pinch | | |

| Minnesota Hand Skill Test | Before Treatment | After Treatment |
|---------------------------------------|------------------|-----------------|
| Placement with the affected hand (sn) | | |
| Placement bilaterally (sn) | | |

## **Gross Motor Functional Classification System (GMFCS)**

## Level of the participant:



| 1 | CHILDHOOD HEALTH ASSESSMENT QUESTIONNAIRE | | | | | |
|---|---|---|---|---|---|---|
| 2 | | | | | | |
| | In this section we are interested in learning how your child's illness affects his/her ability to function in daily life. Please feel free to | | | | | |
| | add any comments on the back of this page. In the following questions, please check the one response which best describes your | | | | | |
| | child's usual activities (averaged over an entire day) OVER THE PAST WEEK, ONLY NOTE THOSE DIFFICULTIES OR | | | | | |
| | LIMITATIONS WHICH ARE DUE TO ILLNESS. If most children at your child's age are not expected to do a certain activity, | | | | | |
| | please mark it as "Not Applicable". For example, if your child has difficulty in doing a certain activity or is unable to do it | | | | | |
| | because he/she is too young but not because he/she is RESTRICTED BY ILLNESS, please mark it as "NOT Applicable". | | | | | |
| | because iterate is too young out my because iterate is to | i i i i i i i i i i i i i i i i i i i | 11.1.1. (1.3.3, р | case mark it | аз пот др | incapit . |
| 3 | | Without | With | With | UNABLE | Not |
| | | ANY | SOME | MUCH | To do | Applicable |
| | | Difficulty | Difficulty | Difficulty | | |
| 4 | DRESSING & GROOMING | | | | | |
| 5 | Is your child able to: | _ | _ | _ | _ | _ |
| 6 | - Dress, including tying shoelaces and doing buttons? | | | | | |
| 7 | - Shampoo his/her hair? | | | | | |
| 8 | Remove socks? | | | | ŏ | ŏ |
| 9 | - Cut fingernails? | | | | | |
| 10 | ARISING | | | | | |
| | Is your child able to: | | | | | |
| 12 | | | | | | |
| 13 | Get in and out of bed or stand up in a crib? | | | | | |
| 14 | EATING | | | | | |
| | Is your child able to: | | | | | |
| 16 | - Cut his/her own meat?<br>- Lift up a cup or glass to mouth? | H | H | H | Н | Н |
| 18 | | ă | ŏ | ŏ | ŏ | ŏ |
| 19 | WALKING Is your child able to: | | | | | |
| 21 | - Walk outdoors on flat ground? | | | | | |
| 22 | - Climb up five steps? | | | | | |
| 23 | * Please check any AIDS or DEVICES that your child us | ually uses for an | y of the above | e activities: | | |
| 24 | Comp | ☐ Davisse | used for descrip | no (button book | l. minnon mult | Ione |
| 24 | - Cane | | shoe horn, etc. | ng (button hoo<br>) | k, zipper pull, | iong- |
| 25 | - Walker | <ul> <li>Built up</li> </ul> | pencil or speci | al utensils | | |
| 26 | Crutches | Special of | or built up chai<br>pecify: | г | | |
| 27 | - Wheelchair | Other (S | pecify: | | | ) 🗆 |
| 28 | * Please check any categories for which your child usual | ly needs help fro | m another per | rson BECAUS | E OF ILLNE | SS: |
| | Position and Consolina | □ materi | | | | |
| 29<br>30 | - Dressing and Grooming<br>- Arising | - Eating - Walking | | | | Н |
| 20 | Arrang | - waiking | | | | |

| 31 | | Without<br>ANY<br>Difficulty | With<br>SOME<br>Difficulty | With<br>MUCH<br>Difficulty | UNABLE<br>To do | Not<br>Applicable |
|---|---|---|---|---|---|---|
| 32 | HYGIENE | | | | | |
| | Is your child able to: | | | | | |
| | Wash and dry entire body? | | | | | |
| 35 | Take a tub bath (get in and out of tub)? | | | | | |
| | Get on and off the toilet or potty chair? | | | | | |
| 37 | | H | H | H | H | H |
| 38 | - Comb/brush hair? | | | | | |
| 39 | REACH | | | | | |
| | Is your child able to: | | | | | |
| | Reach and get down a heavy object such as a large game or | | | | | |
| | books from just above his/her head? | _ | _ | _ | _ | _ |
| 42 | Bend down to pick up clothing or a piece of paper from the | | | | | |
| 43 | floor? | | | | | |
| 43 | Pull on a sweater over his/her head? Turn neck to look back over shoulder? | H | H | H | Н | H |
| • | Turn neck to rook back over shoulder: | | | | | |
| 45 | GRIP | | | | | |
| 46 | Is your child able to: | _ | _ | _ | _ | _ |
| 47 | | | | | | |
| | Open car doors? | Н | Н | H | Н | Н |
| | Open jars which have been previously opened? | H | Н | H | H | H |
| 50<br>51 | - Turn faucets on and off?<br>- Push open a door when he/she has to turn a door knob? | H | H | H | H | Н |
| | That open a door when he are has to turn a door know. | | | _ | | |
| 52 | ACTIVITIES | | | | | |
| | Is your child able to: | | | | | |
| | Run errands and shop? | Н | Н | - 4 | Н | Н |
| | - Get in and out of a car or toy car or school bus?<br>- Ride bike or tricycle? | H | H | H | H | H |
| | Do household chores (e.g. wash dishes, take out trash, | ň | П | Б | ŏ | ŏ |
| | vacuuming, yardwork, make bed, clean room)? | | | | | |
| 58 | Run and play? | | | | | |
| | Please check any AIDS or DEVICES that your child usual<br>Raised toilet seat | | • | activities: | | |
| 61 | Bathtub seat | - Bathtub | oar<br>ndled appliance | es for reach | | H |
| | Jar opener (for jars previously opened) | | ndled appliance | | | ŏ |
| | | | | | | _ |
| | Please check any categories for which your child usually i | | | | E OF ILLNE | SS: |
| | - Hygiene | | and opening to<br>and chores | hings | | H |
| 63 | - Reach | - Errands | and chores | | | |
| 66 | PAIN: We are also interested in learning whether or not your c | hild has been a | iffected by pair | because of his | or her illness | |
| | How much pain do you think your child has had because of his | | | | | |
| | Place a mark on the line below, to indicate the severity of the p | ain | | | | |
| | No pole (0.1 | | Lines | Ioma con con cont | | |
| 67 | No pain 0 | | 100 \ | ery severe pan | n | |
| 68 | GLOBAL EVALUATION: Considering all the ways that arth | ritis affects vo | ur child, rate be | ow he/she is do | ing by placing | a single |
| | mark on the line below. | Jon and Lines Jon | | | and o' brace mile | , |
| 69 | Very well 0 | | 100 | Very poor | | |